CLINICAL TRIAL: NCT02186860
Title: Treatment of Chemotherapy Resistant or Refractory Acute Lymphoblastic Leukemia by Chimeric Antigen Receptor (CAR)-Modified T Cells
Brief Title: Chimeric Antigen Receptor (CAR)-Modified T Cell Therapy in Treating Patients With Acute Lymphoblastic Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 307-CTC-CAR T
Record Dates: First submitted 2014-07-08; First posted 2014-07-10 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CAR-T cells (Experimental): Targeting CD19
  Interventions: Biological: CAR-T cells

INTERVENTIONS:
Biological: CAR-T cells — Given IV

SUMMARY:
Traditional standard treatments of B cell acute lymphoblastic leukemia is not perfect for fighting cancer. Many people do not respond to the standard treatments of ALL. One possible treatment is chimeric antigen receptor (CAR) modified T cell infusions. This study aims to evaluate the safety and efficacy of novel CARTs (targeting CD19) in the treatment of refractory or recurrent ALL.The investigators start Phase I study aimed to chemotherapy resistant or refractory acute lymphoblastic leukemia patients. The purpose of this study is to assess the safety and effectiveness of CAR-T cells in patients.

DETAILED DESCRIPTION:
CAR-T has stronger effect of anti-tumor capacity. While people have been able to control the clinical complications now, so conducting CAR-T clinical trials has a strong demand and value. This study aims to evaluate the safety and efficacy of CD19-CART in treating refractory or recurrent ALL.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years
* Patients with Cluster of Differentiation 19 (CD19) positive B cell malignancies as confirmed by flow cytometry
* Refractory or relapsed B cell-acute lymphoblastic leukemia
* No available curative treatment options (such as hematopoietic stem cell transplantation)
* Stage III-IV disease
* Creatinine < 2.5 mg/dl
* Aspartate transaminase-alanine transaminase ratio < 3x normal
* Bilirubin < 2.0 mg/dl
* Karnofsky performance status >= 60
* Expected survival time > 3 months
* Adequate venous access for apheresis
* Ability to understand and provide informed consent

Exclusion Criteria:

* Pregnant or lactating women
* Patients requiring T cell immunosuppressive therapy
* Active central nervous system leukemia
* Any concurrent active malignancies
* Patients with a history of a seizure disorder or cardiac disorder
* Patients with human immunodeficiency virus, hepatitis B or C infection
* Uncontrolled active infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events | 8 weeks
  To evaluate the safety of CAR-T cells in adult patients with B-acute lymphoblastic leukemia

SECONDARY OUTCOMES:
Clinical responses to third generation CAR-T cells | 2 years
  To assess the anti-leukemic effect of CAR-T cells in adult patients with B cell-acute lymphoblastic leukemia

CONTACTS AND LOCATIONS:
Overall Officials: Liangding Hu, M.D., Principal Investigator — Affiliated Hospital to Academy of Military Medical Sciences
Locations (1):
- Department of Hematopoietic Stem Cell Transplantation, Beijing, China

REFERENCES:
- [Derived] Tang XY, Sun Y, Zhang A, Hu GL, Cao W, Wang DH, Zhang B, Chen H. Third-generation CD28/4-1BB chimeric antigen receptor T cells for chemotherapy relapsed or refractory acute lymphoblastic leukaemia: a non-randomised, open-label phase I trial protocol. BMJ Open. 2016 Dec 30;6(12):e013904. doi: 10.1136/bmjopen-2016-013904. PMID 28039295